CLINICAL TRIAL: NCT06080919
Title: Plaque Modification And Impact On Microcirculatory Territory After Drug-Coated Balloon Percutaneous Coronary Intervention.
Brief Title: Plaque Modification And Impact On Microcirculatory Territory After Drug-Coated Balloon Percutaneous Coronary Intervention (PLAMI).
Acronym: PLAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Jorge Sanz Sanchez, Principal Investigator, Hospital Universitario La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 523
Record Dates: First submitted 2022-09-22; First posted 2023-10-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Drug Coated-balloon; Intravascular Ultrasound; Plaque Modification; Percutaneous Coronary Intervention; Microvascular Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The study will be an investigator-initiated, single-arm, open-label, pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCB-PCI (Experimental): Patients with coronary artery disease undergoing percutaneous coronary intervention will undergo DCB-PCI under IVUS guidance and angio-derived coronary phisiology assessment. Angiographic follow-up with IVUS evaluation will be performed 3 months after the index procedure.
  Interventions: Device: Drug coated-balloon percutaneous coronary intervention.; Device: Angiography-derived coronary physiology (IMRangio)

INTERVENTIONS:
Device: Drug coated-balloon percutaneous coronary intervention. — Patients will undergo DCB-PCI under IVUS guidance (OpticrossTMHD 60 MHz). Target lesion will be predilated with semi-compliant balloons or non-compliant balloons.The lesion will be then treated with DCB with a reference vessel diameter/balloon diameter ratio of 1.
Device: Angiography-derived coronary physiology (IMRangio) — Angiography-derived coronary physiology will be assessed after the procedure using Angio Plus software (Pulse Medical Imaging Technology, Shanghai, China). The angiography images will be used to obtain the IMRangio values, prior and post to DCB-PCI

SUMMARY:
Coronary artery disease (CAD) is one of the most common causes of mortality worldwide. Despite drug eluting stents (DES) are the most common treatment strategy, drug-coated balloons (DCB) represent an appealing alternative to DES as they eliminate the risk of stent thrombosis and do not leave any type of metallic structure in the vessel wall. However, the evidence of the vessel wall healing processes, plaque remodeling, plaque composition and impact on coronary microcirculation after PCI with DCB have not yet been characterized.

The purpose of this study is to assess the changes in percentage atheroma volume evaluated by intravascular ultrasound (IVUS) in patients undergoing DCB-PCI.

DETAILED DESCRIPTION:
The study will be an investigator-initiated, single-arm, open-label, pilot study in patients undergoing PCI with DCB for the novo lesion.

Because of the exploratory nature of this study, no formal sample size calculation is required. On the basis of previous pilot studies with similar designs, a sample of 30 lesions is planned to be evaluated.

After being informed about the study and the potential risks, all patients meeting all the inclusion criteria and none of exclusion criteria will give written informed consent. Patients will go DCB-PCI. IVUS will be evaluated prior to PCI-DCB, immediately after and at 3-month follow-up. Angiography-derived coronary physiology will be assessed after the procedure using Angio Plus software (Pulse Medical Imaging Technology, Shanghai, China). The angiography images will be used to obtain the IMRangio values, prior, post to DCB-PCI and 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with coronary artery disease undergoing percutaneous coronary intervention with DCB.

Exclusion Criteria:

* Aged < 18 years.
* Cardiogenic shock.
* ST-segment elevation myocardial infarction.
* Use of mechanical circulatory support.
* Chronic total occlusions, bifurcation lesions, left main coronary artery disease, severe calcified lesions, graft interventions and in-stent restenosis.
* Inability to provide informed consent.
* Unable to understand and follow study-related instructions or unable to comply with study protocol.
* Currently participating in another trial.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in percentage atheroma volume evaluated by intravascular ultrasound (IVUS) from baseline at 3 month follow-up. | Baseline to 3 month follow-up.

SECONDARY OUTCOMES:
Percentage of minimum lumen change baseline to 3 month follow-up. | Baseline to 3 month follow-up.
Percentage of plaque burden change baseline to 3 month follow-up. | Baseline to 3 month follow-up.
Rate of IMRangio change from baseline to post DCB-PCI | Baseline to post DCB-PCI
Rate of IMRangio change from post DCB-PCI to 3 month follow-up | Post DCB-PCI to 3 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data would be shared under appropriate request

REFERENCES:
- [Background] Stefanini GG, Alfonso F, Barbato E, Byrne RA, Capodanno D, Colleran R, Escaned J, Giacoppo D, Kunadian V, Lansky A, Mehilli J, Neumann FJ, Regazzoli D, Sanz-Sanchez J, Wijns W, Baumbach A. Management of myocardial revascularisation failure: an expert consensus document of the EAPCI. EuroIntervention. 2020 Dec 4;16(11):e875-e890. doi: 10.4244/EIJ-D-20-00487. PMID 32597391
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Sanz Sanchez J, Chiarito M, Cortese B, Moretti A, Pagnotta P, Reimers B, Stefanini GG, Ferrante G. Drug-Coated balloons vs drug-eluting stents for the treatment of small coronary artery disease: A meta-analysis of randomized trials. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):66-75. doi: 10.1002/ccd.29111. Epub 2020 Jun 27. PMID 32592437
- [Background] Xu J, Lo S. Fundamentals and role of intravascular ultrasound in percutaneous coronary intervention. Cardiovasc Diagn Ther. 2020 Oct;10(5):1358-1370. doi: 10.21037/cdt.2020.01.15. PMID 33224762
- [Derived] Sorolla Romero JA, Teira Calderon A, Vilchez Tschischke JP, Aguar Carrascosa P, Ten Morro F, Andres Lalaguna L, Martinez Dolz L, Diez Gil JL, Garcia-Garcia HM, Sanz Sanchez J. [Plaque modification and impact on the microcirculation territory after drug-coated balloon angioplasty. The PLAMI study design]. REC Interv Cardiol. 2024 Mar 4;6(2):83-88. doi: 10.24875/RECIC.M23000438. eCollection 2024 Apr-Jun. PMID 40416350